CLINICAL TRIAL: NCT04494711
Title: A Multi-phased Technology Integrated Physical Literacy Program Targeting Adults With Multimorbidity. A Knowledge Translation Project
Brief Title: Physical Literacy and Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Julie Richardson (Other)
Collaborators: McMaster University (Other)
Responsible Party: Sponsor-Investigator, Julie Richardson, Professor and Assistant Dean School of Rehabilitation Science, McMaster University
Organization: McMaster University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: McMaster University
Record Dates: First submitted 2020-07-28; First posted 2020-07-31 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Chronic Conditions, Multiple; Aging; Mobility Limitation
Keywords: Adults; physical function; physical literacy
MeSH Terms: conditions — Multiple Chronic Conditions; Mobility Limitation

STUDY DESIGN:
Intervention Model Description: Mixed Methods
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical functional literacy (Experimental): 5 week physical literacy program for adults with multiple chronic conditions
  Interventions: Behavioral: Physical Functional Literacy for Adults

INTERVENTIONS:
Behavioral: Physical Functional Literacy for Adults — A 5 week physical literacy for program focused on virtual knowledge translation strategies to improve function and mobility for adults with multiple chronic conditions. This is a population -based approach to rehabilitation

SUMMARY:
With the aging population, the prevalence of chronic conditions continues to rise, affecting 1/3 of Canadians. The promotion of physical literacy, defined as "the motivation, confidence, physical competence and knowledge, to take responsibility for engagement in physical activity for life", has emerged as a promising strategy to increase movement for children. However, little is known about how physical literacy can impact aging adults. A working definition of physical literacy for adults focusing on mobility, function and self-monitoring provides opportunity to guide public health programs in addressing the rehabilitation needs of persons living with multiple chronic conditions.

DETAILED DESCRIPTION:
The objectives of this three stage mixed methods study is to:

1. Develop a new physical literacy framework, with the help of health professionals and end-users that promotes optimal physical functioning for adults.
2. Develop a population-based health intervention using rehabilitation strategies that are delivered virtually to increase physical literacy for adults.

The first 2 qualitative studies will be used to inform the third quantitative intervention.

First, an on-line consensus approach with physiotherapy leaders, rehabilitation researchers and public health experts will be used to identify a new physical literacy framework as it relates to adults.

Second, virtual semi-structured interviews with working adults who are living with 2 or more chronic conditions will determine how aging adults frame physical literacy in their life, specifically with the management of chronic conditions.

Lastly, working adults with 2 or more chronic conditions will participate in a 5-week physical literacy program. Multifaceted knowledge translation strategies including; "walk and talk" with a neighbour or friend, podcasts and on-line mobility challenges will be utilized.

It is anticipated the intervention will improve important physical literacy outcomes such as; physical competence, function, mobility, motivation, awareness, and self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be screened by the primary researcher for the following inclusion criteria:

  1. Diagnosed from a physician with 2 or more chronic conditions and have lived with the conditions for ≥1 year
  2. Able to speak English
  3. Employed full time as a teacher in the Hamilton-Wentworth School Board, Ontario between the ages of 45 and 65 years.
  4. Describe themselves as moderately physically active or inactive over the past 12 months

Exclusion Criteria:

* Advised by physician not to participate in physical activity

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Physical Function at Baseline (Week 1) | Week 1
  The Patient Specific Functional Scale is a patient-reported questionnaire that asks participants to identify up to 5 important activities they are having difficulty with because of their health problem, and to rate their ability to perform those activities on a scale of 0 (unable to perform the activity) to 10 (able to perform the activity like they always have).
Change in Physical Function from Week 1 | Week 5
  The Patient Specific Functional Scale is a patient-reported questionnaire that asks participants to identify up to 5 important activities they are having difficulty with because of their health problem, and to rate their ability to perform those activities on a scale of 0 (unable to perform the activity) to 10 (able to perform the activity like they always have).
Mobility Survey at Baseline (Week 1) | Week 1
  Manty Preclinical Disability Scale: Patient report questionnaire has been created from the work by Many (2007). Self reported mobility is determined by asking participants to rate their ability to walk 2.0 km, walk 0.5 km and climb up 1 flight of stairs on a scale of 1 (able to manage without difficulty) to 5 (unable to manage even with help). To identify persons at an early stage of mobility limitation (preclinical mobility limitation), additional questions were posed to participants who reported no task difficulty. The questions concerned the modification of task performance and the alternatives given were resting in the middle of the performance, using an aid, taking support from handrails, having reduced the frequency of performing the task, having slowed down performance of the task, experiencing tiredness when performing the task, or some other change in carrying out the task.
Change in Mobility from Week 1 | Week 5
  Manty Preclinical Disability Scale: Patient report questionnaire has been created from the work by Many (2007). Self reported mobility is determined by asking participants to rate their ability to walk 2.0 km, walk 0.5 km and climb up 1 flight of stairs on a scale of 1 (able to manage without difficulty) to 5 (unable to manage even with help). To identify persons at an early stage of mobility limitation (preclinical mobility limitation), additional questions were posed to participants who reported no task difficulty. The questions concerned the modification of task performance and the alternatives given were resting in the middle of the performance, using an aid, taking support from handrails, having reduced the frequency of performing the task, having slowed down performance of the task, experiencing tiredness when performing the task, or some other change in carrying out the task.
Self-regulation at Baseline (Week 1) | Week 1
  The Health education impact questionnaire (heiQ): A Patient report questionnaire that aims to evaluate eight self-management skills in people with chronic conditions. Consists of 35 items across 7 independent constructs: health-directed activity; positive and active engagement in life; emotional wellbeing; self-monitoring and insight; constructive attitudes and approaches; skill and technique acquisition; social integration and support. Each construct comprises an independent questionnaire. Each construct-specific questionnaire includes 4-6 items rated on a 4-point scale (1 = strongly disagree, 2 = disagree, 3 = agree, 4 = strongly agree). The sum of scores for all items is divided by the number of items; construct scores range between 1 and 4. A higher score indicates better self-management, with the exception of the emotional wellbeing construct for which a lower score means better emotional well being.
Change in Self-regulation from Week 1 | Week 5
  The Health education impact questionnaire (heiQ): A Patient report questionnaire that aims to evaluate eight self-management skills in people with chronic conditions. Consists of 35 items across 7 independent constructs: health-directed activity; positive and active engagement in life; emotional wellbeing; self-monitoring and insight; constructive attitudes and approaches; skill and technique acquisition; social integration and support. Each construct comprises an independent questionnaire. Each construct-specific questionnaire includes 4-6 items rated on a 4-point scale (1 = strongly disagree, 2 = disagree, 3 = agree, 4 = strongly agree). The sum of scores for all items is divided by the number of items; construct scores range between 1 and 4. A higher score indicates better self-management, with the exception of the emotional wellbeing construct for which a lower score means better emotional well being.

SECONDARY OUTCOMES:
Physical Activity at Baseline (Week 1) | Week 1
  International Physical Activity Questionnaire (IPAQ) Long From: The IPAQ is a 27-item self report questionnaire that measures physical activity for adults between the ages of 15 and 69 years. The questionnaire looks at the types of activities, the intensity of physical activity and sitting time that people do as part of their daily lives. This is used to estimate total physical activity in MET-min/week and time spent sitting. There are 5 domains of physical activity within the long version of the IPAQ (job related, transportation, house work/house maintenance/caring for family, recreation/sport/leisure time and time spent sitting.
  Participants are scored as either Low (lowest level of physical activity), Moderate or High physical activity
Change in Physical Activity from week 1 | Week 5
  International Physical Activity Questionnaire (IPAQ) Long From: The IPAQ is a 27-item self report questionnaire that measures physical activity for adults between the ages of 15 and 69 years. The questionnaire looks at the types of activities, the intensity of physical activity and sitting time that people do as part of their daily lives. This is used to estimate total physical activity in MET-min/week and time spent sitting. There are 5 domains of physical activity within the long version of the IPAQ (job related, transportation, house work/house maintenance/caring for family, recreation/sport/leisure time and time spent sitting.
  Participants are scored as either Low (lowest level of physical activity), Moderate or High physical activity
Self-efficacy to manage chronic conditions at Baseline (Week 1) | Week 1
  A 10-point self-efficacy scale to determine participant's confidence in managing their chronic conditions. Participants will be asked to rate how confident they are with self-managing their chronic conditions on a daily basis using a single question on a scale of 1 - 10. Higher values equal greater self-efficacy.
Change in Self-efficacy from week 1 | Week 5
  A 10-point self-efficacy scale to determine participant's confidence in managing their chronic conditions. Participants will be asked to rate how confident they are with self-managing their chronic conditions on a daily basis using a single question on a scale of 1 - 10. Higher values equal greater self-efficacy.
Knowledge and Awareness of health changes that occur with aging Baseline (Week 1) | Week 1
  Participants will be asked to answer 2 open-ended questions related to changes that occur with mobility and physical function with aging. Question 1: Name changes that occur with aging and chronic conditions that affect one's ability to move and get around with ease. Question 2: Name things you can do to improve your health and ability to move around despite living with chronic conditions. Higher scores will be based on the higher number of correct answers.
Change in Awareness level from week 1 | Week 5
  Participants will be asked to answer 2 open-ended questions related to changes that occur with mobility and physical function with aging. Question 1: Name changes that occur with aging and chronic conditions that affect one's ability to move and get around with ease. Question 2: Name things you can do to improve your health and ability to move around despite living with chronic conditions. Higher scores will be based on the higher number of correct answers.
Participant satisfaction of the Physical Literacy program | Week 5
  Participants will be asked to rate their satisfaction of the physical literacy program at the end of the 5 week study period. They will be asked "Overall on a scale of 0 - 10 how would you rate your experience with the physical literacy program?" Higher numbers will equate to a higher satisfaction score.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Richardson, PhD, Principal Investigator — McMaster University
Locations (1):
- Celeste Petrusevski, Hamilton, Canada

IPD SHARING:
Plan to Share IPD: No